CLINICAL TRIAL: NCT06014047
Title: Graft Patency Between the Radial Artery and the No-touch Saphenous Vein in Coronary Artery Bypass Grafting Study (GRAFT-CAB Study)
Brief Title: Radial Artery Versus No-touch Saphenous Vein
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2109
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Touch vein (Experimental): No-touch vein group has two No-touch saphenous vein grafts, anastomose to the right coronary or left coronary system. All patients also acquired LITA-LAD anastomosis to complete the revascularization.
  Interventions: Procedure: No-touch vein graft
- Radial artery (Active Comparator): Radial artery group has one radial artery graft and one conventional saphenous vein graft, anastomose to the right coronary or left coronary system basing on surgeons' decision. All patients also acquired LITA-LAD anastomosis to complete the revascularization.
  Interventions: Procedure: Radial artery graft

INTERVENTIONS:
Procedure: No-touch vein graft — Two No-touch saphenous vein grafts anastomose to the right coronary and left coronary system. All participants also acquired Left intrathoracic artery(LITA)-left anterior decending artery(LAD) anastomosis to complete the revascularization.
  Arms: No-Touch vein
Procedure: Radial artery graft — One radial artery graft and one conventional saphenous vein graft anastomose to the right coronary or left coronary system basing on surgeons' decision. All participants also acquired Left intrathoracic artery(LITA)-left anterior decending artery(LAD) anastomosis to complete the revascularization.
  Arms: Radial artery

SUMMARY:
This study evaluates the short-term and long-term patency of the radial artery and the No-touch vein in patients undergoing isolated on-pump/off-pump coronary artery bypass graft (CABG) surgery. A total of at least 774 patients undergoing isolated on-pump/off-pump CABG will be consecutively recruited from Fuwai Hospital and randomly assigned to receive radial artery or No-touch saphenous vein as their second graft. All participants will be invited for clinical follow-up and 64-slice multislice computed tomography angiography (MSCTA) analysis at 3 months and 12 months post-operatively.

DETAILED DESCRIPTION:
CABG is still the treatment of choice for ischemic heart disease. However, restenosis or occlusion may occur to graft vessels, leading to postoperative myocardial ischemia and subsequent clinical events. Long-term angiographic follow-up demonstrated that vein graft restenosis and occlusion are common among those receiving CABG, with a vein graft patency of less than 50% at 15 years postoperatively.

A novel approach to harvesting the vein is called "No-touch" technique (NT), which can avoid mechanical damage to the vein wall. Previous studies showed that No-touch saphenous vein grafts (NT-SVG) has a 96.3% postoperative graft patency rate at 12 months, compared to 93.5% of conventional saphenous vein grafts (con-SVGs). Thus, the No-touch technique can significantly reduce postoperative graft occlusion. Radial artery(RA) as an arterial material for CABG surgery has a better long-term patency than con-SVG, up to 83% at 10 years. Using radial artery as the second graft for CABG may provide additional clinical benefit. However, the risk of perioperative vasospasm and graft occlusion due to competitive blood flow limit the using of radial artery. Therefore, only the No-touch vein and the radial artery can improve the graft patency. Only one randomized clinical trial(RCT) compared the RA and NT-vein, and this study is limited by irregular post-operative management and small sample size from single center.

This prospective single-center study aims to compare the short-term and long-term graft patency between the No-touch vein and the radial artery. This study will consecutively enroll at least 774 patients undergoing isolated on-pump/off-pump CABG. After obtaining informed written consent, participants will be randomly allocated to either the No-touch or the radial artery group. At baseline, participants will be interviewed to collect detailed information about on demographics, socioeconomic status, cardiovascular risk factors, clinical characteristics, treatments, in-hospital outcomes, general and disease-specific quality of life, function and mental status. During the follow-ups, the investigators will collect information about clinical outcomes events, long-term treatments, function, quality of life, symptoms, and medical care during the recovery period. All participants will be invited for 64-slice multi-slice computed tomography angiography (MSCTA) analysis at 3 months and 12 months post-operatively for graft patency evaluation.

The data adjudicators and computed tomography(CT) reviewers will be blinded to the study. Due to the nature of this study, the operating surgeons, anesthetists and other operative room staff will not be blind in this study. Owing to the use of radial artery need approved by the participant, so participants will also not be blind in this study,

By comparing the short-term and long-term graft patency between the No-touch vein and radial artery groups, this study will contribute major evidence of the possible superiority between two different grafts, so as to improve patient outcomes after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* First time undergo isolated CABG surgery
* Severe three-vessel disease (Left anterior decending artery, Left circumflex artery, Right coronoary artery lesion with more than 75% stenosis)

Exclusion Criteria:

* Urgent or Redo CABG surgery
* Concomitant cardiac or vascular procedures (i.e. valve repair or replacement, Morrow procedure)
* A positive Allen test, radial artery plaque on ultrasound or a history of vasculitis or Raynaud's syndrome
* Varicose great saphenous vein or venous tortuosity and judged as can not be used in operation by surgeons
* Known allergy to radiographic contrast media
* Planed endarterectomy of coronary artery before surgery
* Malignant tumor or other severe systemic diseases
* Combined with other irreversible organ failures
* Contraindications for dual antiplatelet therapy, such as active gastroduodenal ulcer
* Participant of other ongoing clinical trials in 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of graft patency | 12 months after procedure
  All participants will be invited to return to their operating hospitals for 64-slice multi-slice computed tomography angiography to determine patencies of the graft vessels.

SECONDARY OUTCOMES:
Prevalence of graft patency | 3 months, 3 years and 5 years after procedure
  All participants will be invited to return to their operating hospitals for 64-slice multi-slice computed tomography angiography to determine patencies of the graft vessels.
Overall major adverse cardiac or cerebrovascular events (MACCE) rate | 3 months, 12 months, 3 years and 5 years after procedure
  MACCE includes death, myocardial infarction, stroke and/or repeat revascularization
Cardiac death | 3 months, 12 months, 3 years and 5 years after procedure
  Death from any heart disease
Documented non-lethal myocardial infarction | 3 months, 12 months, 3 years and 5 years after procedure
  Myocardial infarction is defined according to the most recent guideline
Stroke | 3 months, 12 months, 3 years and 5 years after procedure
  An acute symptomatic episode of focal or global neurological dysfunction caused by brain, spinal, or retinal vascular injury as a result of hemorrhage or infarction
Target lesion revascularization | 3 months, 12 months, 3 years and 5 years after procedure
  CABG or percutaneous coronary intervention
Recurrence of Angina | 3 months, 12 months, 3 years and 5 years after procedure
  Recurrence of Angina

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academay of Medical Science and National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tian M, Wang X, Sun H, Feng W, Song Y, Lu F, Wang L, Wang Y, Xu B, Wang H, Liu S, Liu Z, Chen Y, Miao Q, Su P, Yang Y, Guo S, Lu B, Sun Z, Liu K, Zhang C, Wu Y, Xu H, Zhao W, Han C, Zhou X, Wang E, Huo X, Hu S. No-Touch Versus Conventional Vein Harvesting Techniques at 12 Months After Coronary Artery Bypass Grafting Surgery: Multicenter Randomized, Controlled Trial. Circulation. 2021 Oct 5;144(14):1120-1129. doi: 10.1161/CIRCULATIONAHA.121.055525. Epub 2021 Sep 13. PMID 34510911
- [Result] Nappi F, Bellomo F, Nappi P, Chello C, Iervolino A, Chello M, Acar C. The Use of Radial Artery for CABG: An Update. Biomed Res Int. 2021 Apr 7;2021:5528006. doi: 10.1155/2021/5528006. eCollection 2021. PMID 33928147
- [Derived] Zhang F, Tian M, Wang X, Zhang H, Zhou X, Liu R, Liu R, Jin Z, Zhang C, Wang X. Rationale and design of a single-center randomized trial to compare the graft patency between the radial artery and the no-touch saphenous vein in coronary artery bypass grafting surgery (GRAFT-CAB Study). Am Heart J. 2024 Aug;274:46-53. doi: 10.1016/j.ahj.2024.05.001. Epub 2024 May 6. PMID 38710379